CLINICAL TRIAL: NCT03324009
Title: Development of a Two-stage Cervical Cancer Screening Algorithm for Botswana
Brief Title: 2-stage Cervical Cancer Screening in Botswana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Rebecca Luckett, Instructor in Obstetrics, Gynecology and Reproductive Biology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017P000388; 5P30AI060354-14 (NIH)
Record Dates: First submitted 2017-10-12; First posted 2017-10-27 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Cervical Cancer; HIV/AIDS
MeSH Terms: conditions — Uterine Cervical Neoplasms; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 2-stage screen (Experimental): All patients will be enrolled in the two-stage cervical cancer screening protocol
  Interventions: Diagnostic Test: 2-stage screen

INTERVENTIONS:
Diagnostic Test: 2-stage screen — Pap smear is currently the standard of care for cervical cancer screening in Botswana. In this study, participants will undergo HPV DNA testing at the time of Pap smear collection. If HPV DNA test is positive, they will be referred for colposcopy. Patients who have an HPV negative test but positive Pap smear will be referred for colposcopy per Botswana cervical cancer screening guidelines.

SUMMARY:
Cervical cancer is the leading cause of cancer death among women in Botswana. The burden of cervical cancer is largely related to the high prevalence of HIV in Botswana (22%), as HIV is known to be a significant risk factor for cervical cancer. Cervical cancer screening is life-saving and has been shown to reduce cervical cancer incidence in multiple settings. Yet, there is no consensus on appropriate screening algorithms for women living with HIV, across resource settings. Botswana is in a unique position, relative to its neighbors in Sub-Saharan Africa, in that there exists capacity for advanced screening modalities, including primary high risk human papilloma virus (hrHPV) testing and cytology-based screening. To address this issue, this study seeks to evaluate two-stage cervical cancer screening algorithms for women living with HIV in Botswana using hrHPV testing. The protocols include hrHPV testing followed by Pap Smear evaluation, VIA and colposcopy. These same participants will be invited back at one-year for cervical cancer screening using hrHPV testing (followed by triage testing) in order to inform guidelines on the frequency of HPV testing in women living with HIV. The evidence generated will be critical to guiding cervical cancer screening in HIV-infected women across resource settings.

DETAILED DESCRIPTION:
Cervical cancer screening programs vary across settings and there is no clear guidance for effective screening programs for HIV-positive women. Evaluating the performance of algorithms that include human papillomavirus (HPV) DNA testing as first stage screening in high HIV prevalence settings like Botswana is essential for establishing an evidence-based strategy for cervical cancer screening in HIV-positive women.

This study seeks to evaluate the performance of two-stage cervical cancer screening algorithms using primary HPV testing in women living with HIV in Botswana. Second stage screening modalities include Papanicolaou (Pap) smear, visual inspection with acetic acid (VIA) and colposcopy.

The study will enroll 300 HIV positive women. For all 300 participants, gynecologic speculum exam will be performed and provider-collected cervical swabs will be collected for HPV testing and Pap smear preparation. HPV testing will be performed with either the commercially-available Cepheid Xpert® HPV Assay or a high throughput PCR platform. Pap smear will be prepared using standard technique at the site of collection.

Participants who test HPV-negative will have their Pap smear sent to the National Health Lab (NHL) for staining and pathologist evaluation. If the Pap smear is abnormal, they will be referred to colposcopy per current Botswana Cervical Cancer Prevention Guidelines.

Participants who test HPV-positive will also have their Pap smear reviewed, and will also be asked to return for colposcopy and will undergo further diagnosis and treatment for cervical cancer per national guidelines. At the colposcopy visit, a trained nurse will conduct VIA using the Botswana standard protocol. After application of acetic acid to the cervix, the nurse will record visual results as positive or negative. If VIA is positive based on assessment of the lesion(s), the nurse will record a recommendation for either cryotherapy or loop electrosurgical excision procedure (LEEP). Since all of these HPV-positive participants will undergo colposcopy, the participants will not be informed of the VIA results, as neither cryotherapy nor LEEP will be administered based on the VIA results. Rather, the participants will proceed to colposcopy and results of colposcopy will determine further diagnosis and treatment. This design enables us to assess the utility of the two-stage algorithms while providing the highest-quality follow-up to cervical cancer screening abnormalities in Botswana.

These same participants will be invited back at one-year for repeat cervical cancer screening using the same screening methods as at baseline. The data will inform guidelines on the frequency of hrHPV testing in women living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* ≥25 years of age
* HIV-positive
* Competent to understand study procedures and give informed consent.

Exclusion Criteria:

* Currently pregnant
* Currently menstruating or having persistent vaginal discharge
* Previous hysterectomy
* Previous diagnosis of cervical cancer

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Performance of HPV-Pap screening algorithm | 2 months
  Measurement of the sensitivity, specificity and positive predictive value of Pap smear in predicting cervical precancer and cancer in HPV positive, HIV positive women.
Performance of HPV-VIA screening algorithm | 2 months
  Measurement of the sensitivity, specificity and positive predictive value of VIA in predicting cervical precancer and cancer in HPV positive, HIV positive women.
Performance of HPV-Colposcopy screening algorithm | 6 months
  Measurement of the sensitivity, specificity and positive predictive value of Colposcopy in predicting cervical precancer and cancer in HPV positive, HIV positive women.
Incident and persistent HPV infection at one-year follow-up | 18 months
Incidence, persistence and progression of histopathologic abnormality at one-year follow-up | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Luckett, MD MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Grover S, Raesima M, Bvochora-Nsingo M, Chiyapo SP, Balang D, Tapela N, Balogun O, Kayembe MK, Russell AH, Monare B, Tanyala S, Bhat J, Thipe K, Nchunga M, Mayisela S, Kizito B, Ho-Foster A, Gaolebale BE, Gaolebale PA, Efstathiou JA, Dryden-Peterson S, Zetola N, Hahn SM, Robertson ES, Lin LL, Morroni C, Ramogola-Masire D. Cervical Cancer in Botswana: Current State and Future Steps for Screening and Treatment Programs. Front Oncol. 2015 Nov 3;5:239. doi: 10.3389/fonc.2015.00239. eCollection 2015. PMID 26579491
- [Background] Ellerbrock TV, Chiasson MA, Bush TJ, Sun XW, Sawo D, Brudney K, Wright TC Jr. Incidence of cervical squamous intraepithelial lesions in HIV-infected women. JAMA. 2000 Feb 23;283(8):1031-7. doi: 10.1001/jama.283.8.1031. PMID 10697063
- [Background] Chin KM, Sidhu JS, Janssen RS, Weber JT. Invasive cervical cancer in human immunodeficiency virus-infected and uninfected hospital patients. Obstet Gynecol. 1998 Jul;92(1):83-7. doi: 10.1016/s0029-7844(98)00140-9. PMID 9649099
- [Background] Peirson L, Fitzpatrick-Lewis D, Ciliska D, Warren R. Screening for cervical cancer: a systematic review and meta-analysis. Syst Rev. 2013 May 24;2:35. doi: 10.1186/2046-4053-2-35. PMID 23706117
- [Background] Gibb RK, Martens MG. The impact of liquid-based cytology in decreasing the incidence of cervical cancer. Rev Obstet Gynecol. 2011;4(Suppl 1):S2-S11. PMID 21617785
- [Background] de Martel C, Ferlay J, Franceschi S, Vignat J, Bray F, Forman D, Plummer M. Global burden of cancers attributable to infections in 2008: a review and synthetic analysis. Lancet Oncol. 2012 Jun;13(6):607-15. doi: 10.1016/S1470-2045(12)70137-7. Epub 2012 May 9. PMID 22575588
- [Background] McCredie MR, Sharples KJ, Paul C, Baranyai J, Medley G, Jones RW, Skegg DC. Natural history of cervical neoplasia and risk of invasive cancer in women with cervical intraepithelial neoplasia 3: a retrospective cohort study. Lancet Oncol. 2008 May;9(5):425-34. doi: 10.1016/S1470-2045(08)70103-7. Epub 2008 Apr 11. PMID 18407790
- [Background] Wheeler CM. Natural history of human papillomavirus infections, cytologic and histologic abnormalities, and cancer. Obstet Gynecol Clin North Am. 2008 Dec;35(4):519-36; vii. doi: 10.1016/j.ogc.2008.09.006. PMID 19061814
- [Background] Denny LA, Franceschi S, de Sanjose S, Heard I, Moscicki AB, Palefsky J. Human papillomavirus, human immunodeficiency virus and immunosuppression. Vaccine. 2012 Nov 20;30 Suppl 5:F168-74. doi: 10.1016/j.vaccine.2012.06.045. PMID 23199960
- [Background] de Sanjose S, Diaz M, Castellsague X, Clifford G, Bruni L, Munoz N, Bosch FX. Worldwide prevalence and genotype distribution of cervical human papillomavirus DNA in women with normal cytology: a meta-analysis. Lancet Infect Dis. 2007 Jul;7(7):453-9. doi: 10.1016/S1473-3099(07)70158-5. PMID 17597569
- [Background] Banura C, Franceschi S, Doorn LJ, Arslan A, Wabwire-Mangen F, Mbidde EK, Quint W, Weiderpass E. Infection with human papillomavirus and HIV among young women in Kampala, Uganda. J Infect Dis. 2008 Feb 15;197(4):555-62. doi: 10.1086/526792. PMID 18237268
- [Background] Dunne EF, Unger ER, Sternberg M, McQuillan G, Swan DC, Patel SS, Markowitz LE. Prevalence of HPV infection among females in the United States. JAMA. 2007 Feb 28;297(8):813-9. doi: 10.1001/jama.297.8.813. PMID 17327523
- [Background] Clifford GM, Smith JS, Plummer M, Munoz N, Franceschi S. Human papillomavirus types in invasive cervical cancer worldwide: a meta-analysis. Br J Cancer. 2003 Jan 13;88(1):63-73. doi: 10.1038/sj.bjc.6600688. PMID 12556961
- [Background] Smith JS, Lindsay L, Hoots B, Keys J, Franceschi S, Winer R, Clifford GM. Human papillomavirus type distribution in invasive cervical cancer and high-grade cervical lesions: a meta-analysis update. Int J Cancer. 2007 Aug 1;121(3):621-32. doi: 10.1002/ijc.22527. PMID 17405118
- [Background] de Sanjose S, Quint WG, Alemany L, Geraets DT, Klaustermeier JE, Lloveras B, Tous S, Felix A, Bravo LE, Shin HR, Vallejos CS, de Ruiz PA, Lima MA, Guimera N, Clavero O, Alejo M, Llombart-Bosch A, Cheng-Yang C, Tatti SA, Kasamatsu E, Iljazovic E, Odida M, Prado R, Seoud M, Grce M, Usubutun A, Jain A, Suarez GA, Lombardi LE, Banjo A, Menendez C, Domingo EJ, Velasco J, Nessa A, Chichareon SC, Qiao YL, Lerma E, Garland SM, Sasagawa T, Ferrera A, Hammouda D, Mariani L, Pelayo A, Steiner I, Oliva E, Meijer CJ, Al-Jassar WF, Cruz E, Wright TC, Puras A, Llave CL, Tzardi M, Agorastos T, Garcia-Barriola V, Clavel C, Ordi J, Andujar M, Castellsague X, Sanchez GI, Nowakowski AM, Bornstein J, Munoz N, Bosch FX; Retrospective International Survey and HPV Time Trends Study Group. Human papillomavirus genotype attribution in invasive cervical cancer: a retrospective cross-sectional worldwide study. Lancet Oncol. 2010 Nov;11(11):1048-56. doi: 10.1016/S1470-2045(10)70230-8. Epub 2010 Oct 15. PMID 20952254
- [Background] Ramogola-Masire D, McGrath CM, Barnhart KT, Friedman HM, Zetola NM. Subtype distribution of human papillomavirus in HIV-infected women with cervical intraepithelial neoplasia stages 2 and 3 in Botswana. Int J Gynecol Pathol. 2011 Nov;30(6):591-6. doi: 10.1097/PGP.0b013e31821bf2a6. PMID 21979597
- [Background] Macleod IJ, O'Donnell B, Moyo S, Lockman S, Shapiro RL, Kayembe M, van Widenfelt E, Makhema J, Essex M, Wester C. Prevalence of human papillomavirus genotypes and associated cervical squamous intraepithelial lesions in HIV-infected women in Botswana. J Med Virol. 2011 Oct;83(10):1689-95. doi: 10.1002/jmv.22178. PMID 21837784
- [Background] Ginsburg O, Badwe R, Boyle P, Derricks G, Dare A, Evans T, Eniu A, Jimenez J, Kutluk T, Lopes G, Mohammed SI, Qiao YL, Rashid SF, Summers D, Sarfati D, Temmerman M, Trimble EL, Padela AI, Aggarwal A, Sullivan R. Changing global policy to deliver safe, equitable, and affordable care for women's cancers. Lancet. 2017 Feb 25;389(10071):871-880. doi: 10.1016/S0140-6736(16)31393-9. Epub 2016 Nov 1. PMID 27814964
- [Background] Lazcano-Ponce E, Lorincz AT, Cruz-Valdez A, Salmeron J, Uribe P, Velasco-Mondragon E, Nevarez PH, Acosta RD, Hernandez-Avila M. Self-collection of vaginal specimens for human papillomavirus testing in cervical cancer prevention (MARCH): a community-based randomised controlled trial. Lancet. 2011 Nov 26;378(9806):1868-73. doi: 10.1016/S0140-6736(11)61522-5. Epub 2011 Nov 1. PMID 22051739
- [Background] Chatzistamatiou K, Moysiadis T, Angelis E, Kaufmann A, Skenderi A, Jansen-Duerr P, Lekka I, Kilintzis V, Angelidou S, Katsiki E, Hagemann I, Tsertanidou A, Koch I, Boecher O, Soutschek E, Maglaveras N, Agorastos T. Diagnostic accuracy of high-risk HPV DNA genotyping for primary cervical cancer screening and triage of HPV-positive women, compared to cytology: preliminary results of the PIPAVIR study. Arch Gynecol Obstet. 2017 May;295(5):1247-1257. doi: 10.1007/s00404-017-4324-x. Epub 2017 Mar 23. PMID 28337594
- [Background] Cuzick J, Clavel C, Petry KU, Meijer CJ, Hoyer H, Ratnam S, Szarewski A, Birembaut P, Kulasingam S, Sasieni P, Iftner T. Overview of the European and North American studies on HPV testing in primary cervical cancer screening. Int J Cancer. 2006 Sep 1;119(5):1095-101. doi: 10.1002/ijc.21955. PMID 16586444
- [Background] Jeronimo J, Castle PE, Temin S, Shastri SS. Secondary Prevention of Cervical Cancer: American Society of Clinical Oncology Resource-Stratified Clinical Practice Guideline Summary. J Oncol Pract. 2017 Feb;13(2):129-133. doi: 10.1200/JOP.2016.017889. Epub 2016 Nov 15. No abstract available. PMID 27845871
- [Background] Wright TC Jr, Ellerbrock TV, Chiasson MA, Van Devanter N, Sun XW. Cervical intraepithelial neoplasia in women infected with human immunodeficiency virus: prevalence, risk factors, and validity of Papanicolaou smears. New York Cervical Disease Study. Obstet Gynecol. 1994 Oct;84(4):591-7. PMID 8090399
- [Background] Mustafa RA, Santesso N, Khatib R, Mustafa AA, Wiercioch W, Kehar R, Gandhi S, Chen Y, Cheung A, Hopkins J, Ma B, Lloyd N, Wu D, Broutet N, Schunemann HJ. Systematic reviews and meta-analyses of the accuracy of HPV tests, visual inspection with acetic acid, cytology, and colposcopy. Int J Gynaecol Obstet. 2016 Mar;132(3):259-65. doi: 10.1016/j.ijgo.2015.07.024. Epub 2015 Nov 12. PMID 26851054
- [Background] Arbyn M, Sankaranarayanan R, Muwonge R, Keita N, Dolo A, Mbalawa CG, Nouhou H, Sakande B, Wesley R, Somanathan T, Sharma A, Shastri S, Basu P. Pooled analysis of the accuracy of five cervical cancer screening tests assessed in eleven studies in Africa and India. Int J Cancer. 2008 Jul 1;123(1):153-60. doi: 10.1002/ijc.23489. PMID 18404671
- [Background] Sankaranarayanan R, Esmy PO, Rajkumar R, Muwonge R, Swaminathan R, Shanthakumari S, Fayette JM, Cherian J. Effect of visual screening on cervical cancer incidence and mortality in Tamil Nadu, India: a cluster-randomised trial. Lancet. 2007 Aug 4;370(9585):398-406. doi: 10.1016/S0140-6736(07)61195-7. PMID 17679017
- [Background] Ronco G, Dillner J, Elfstrom KM, Tunesi S, Snijders PJ, Arbyn M, Kitchener H, Segnan N, Gilham C, Giorgi-Rossi P, Berkhof J, Peto J, Meijer CJ; International HPV screening working group. Efficacy of HPV-based screening for prevention of invasive cervical cancer: follow-up of four European randomised controlled trials. Lancet. 2014 Feb 8;383(9916):524-32. doi: 10.1016/S0140-6736(13)62218-7. Epub 2013 Nov 3. PMID 24192252
- [Background] Sankaranarayanan R, Nene BM, Shastri SS, Jayant K, Muwonge R, Budukh AM, Hingmire S, Malvi SG, Thorat R, Kothari A, Chinoy R, Kelkar R, Kane S, Desai S, Keskar VR, Rajeshwarkar R, Panse N, Dinshaw KA. HPV screening for cervical cancer in rural India. N Engl J Med. 2009 Apr 2;360(14):1385-94. doi: 10.1056/NEJMoa0808516. PMID 19339719
- [Background] Denny L, Kuhn L, De Souza M, Pollack AE, Dupree W, Wright TC Jr. Screen-and-treat approaches for cervical cancer prevention in low-resource settings: a randomized controlled trial. JAMA. 2005 Nov 2;294(17):2173-81. doi: 10.1001/jama.294.17.2173. PMID 16264158
- [Background] Denny L, Kuhn L, Hu CC, Tsai WY, Wright TC Jr. Human papillomavirus-based cervical cancer prevention: long-term results of a randomized screening trial. J Natl Cancer Inst. 2010 Oct 20;102(20):1557-67. doi: 10.1093/jnci/djq342. Epub 2010 Sep 30. PMID 20884893
- [Background] Denny LA, Sankaranarayanan R, De Vuyst H, Kim JJ, Adefuye PO, Alemany L, Adewole IF, Awolude OA, Parham G, de Sanjose S, Bosch FX. Recommendations for cervical cancer prevention in sub-saharan Africa. Vaccine. 2013 Dec 29;31 Suppl 5:F73-4. doi: 10.1016/j.vaccine.2012.11.077. No abstract available. PMID 24331750
- [Background] Santesso N, Mustafa RA, Schunemann HJ, Arbyn M, Blumenthal PD, Cain J, Chirenje M, Denny L, De Vuyst H, Eckert LO, Forhan SE, Franco EL, Gage JC, Garcia F, Herrero R, Jeronimo J, Lu ER, Luciani S, Quek SC, Sankaranarayanan R, Tsu V, Broutet N; Guideline Support Group. World Health Organization Guidelines for treatment of cervical intraepithelial neoplasia 2-3 and screen-and-treat strategies to prevent cervical cancer. Int J Gynaecol Obstet. 2016 Mar;132(3):252-8. doi: 10.1016/j.ijgo.2015.07.038. Epub 2015 Dec 14. PMID 26868062
- [Background] Denny L, Kuhn L, Risi L, Richart RM, Pollack A, Lorincz A, Kostecki F, Wright TC Jr. Two-stage cervical cancer screening: an alternative for resource-poor settings. Am J Obstet Gynecol. 2000 Aug;183(2):383-8. doi: 10.1067/mob.2000.105871. PMID 10942474
- [Background] Naucler P, Ryd W, Tornberg S, Strand A, Wadell G, Elfgren K, Radberg T, Strander B, Forslund O, Hansson BG, Hagmar B, Johansson B, Rylander E, Dillner J. Efficacy of HPV DNA testing with cytology triage and/or repeat HPV DNA testing in primary cervical cancer screening. J Natl Cancer Inst. 2009 Jan 21;101(2):88-99. doi: 10.1093/jnci/djn444. Epub 2009 Jan 13. PMID 19141778
- [Background] Bigoni J, Gundar M, Tebeu PM, Bongoe A, Schafer S, Fokom-Domgue J, Catarino R, Tincho EF, Bougel S, Vassilakos P, Petignat P. Cervical cancer screening in sub-Saharan Africa: a randomized trial of VIA versus cytology for triage of HPV-positive women. Int J Cancer. 2015 Jul 1;137(1):127-34. doi: 10.1002/ijc.29353. Epub 2014 Dec 5. PMID 25420434
- [Background] Ramogola-Masire D, de Klerk R, Monare B, Ratshaa B, Friedman HM, Zetola NM. Cervical cancer prevention in HIV-infected women using the "see and treat" approach in Botswana. J Acquir Immune Defic Syndr. 2012 Mar 1;59(3):308-13. doi: 10.1097/QAI.0b013e3182426227. PMID 22134146
- [Background] Kuhn L, Denny L, Pollack A, Lorincz A, Richart RM, Wright TC. Human papillomavirus DNA testing for cervical cancer screening in low-resource settings. J Natl Cancer Inst. 2000 May 17;92(10):818-25. doi: 10.1093/jnci/92.10.818. PMID 10814677
- See also: Worldwide cervical cancer statistics — http://globocan.iarc.fr

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT03324009/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT03324009/ICF_002.pdf